CLINICAL TRIAL: NCT03876665
Title: The Experience of Living With Polycystic Ovary Syndrome in the Military
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); Malcolm Grow Medical Clinics and Surgery Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH#20200123H
Record Dates: First submitted 2019-02-26; First posted 2019-03-15 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Military; Service Women; Active Duty
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Group: Active Duty Air Force, Army and Navy women diagnosed with PCOS.
  Up to three focus groups per service branch will be conducted. Considering attrition for those who may volunteer and not show up for the FG session, the investigators will recruit up to 20 participants per site, with the goal of including a maximum of six participants per FG to maximize individual participation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to understand the experience of living with polycystic ovary syndrome (PCOS) as an active duty Service Woman. As part of a budding research program, this proposed study will lay the groundwork for future intervention studies targeting the management of PCOS in a military population.

DETAILED DESCRIPTION:
Using a qualitative descriptive approach with focus groups (FG) and individual interviews (II), the investigators will seek to describe the experience of living with PCOS as an active duty service woman (ADSW). This method will allow the investigators to obtain a comprehensive summary of living with PCOS in the every day terms of ADSW. The discussion in the (FG) meetings will be an effective way to supply information about what people think, or how they feel, or on the way they act. Advantages of this method include: (a) it can cover a large number of people in one session, (b) it is an efficient way of gaining a large amount of information in a short time, (c) it is comparatively easier to drive or conduct, and (d) it generates an opportunity to collect data from the group interaction, which concentrates on the topic of the researcher's interest [64, 65].

This proposed study will focus on six primary areas of inquiry: (a) experience of receiving PCOS diagnosis (b) symptoms experienced and methods of coping with them, (c) military-specific experience of managing and living with PCOS, (d) access to/availability of information related to PCOS and how they have applied it, (e) experience of support, and (f) present and future concerns about having PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women, active duty or prior (within 5 years) in the Army, Navy, Air Force or Marine Corps
* Diagnosed with PCOS
* 18 years of age or over

Exclusion Criteria:

* Reservist, Coast Guard, women who have separated or retired > 5 years ago

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female specific condition
Study Population: Active duty military women diagnosed with PCOS
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Describe the PCOS experience of active duty service members | through study completion, up to 18 months
  Information from focused groups (FG) discussions and individual interviews (II) will be transcribed, categorized and then organized into themes that describe the experiences of active duty service members
Describe the PCOS experience by branch of service | through study completion, up to 18 months
  Information from focused groups (FG) discussions and individual interviews (II) will be transcribed, categorized and then organized into themes that describe the experiences by branch of service

CONTACTS AND LOCATIONS:
Overall Officials: Dawnkimberly Hopkins, PhD, Principal Investigator — David Grant Medical Center; Leilani Siaki, PhD, Principal Investigator — Madigan Army Medical Center; Abigail Yablonsky, PhD, Principal Investigator — United States Naval Medical Center, San Diego; Angela Phillips, PhD, Principal Investigator — Malcolm Grow Medical Clinics and Surgery Center
Locations (1):
- David Grant Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azziz R, Carmina E, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Futterweit W, Janssen OE, Legro RS, Norman RJ, Taylor AE, Witchel SF; Task Force on the Phenotype of the Polycystic Ovary Syndrome of The Androgen Excess and PCOS Society. The Androgen Excess and PCOS Society criteria for the polycystic ovary syndrome: the complete task force report. Fertil Steril. 2009 Feb;91(2):456-88. doi: 10.1016/j.fertnstert.2008.06.035. Epub 2008 Oct 23. PMID 18950759
- [Background] Yildizhan B, Anik Ilhan G, Pekin T. The impact of insulin resistance on clinical, hormonal and metabolic parameters in lean women with polycystic ovary syndrome. J Obstet Gynaecol. 2016 Oct;36(7):893-896. doi: 10.3109/01443615.2016.1168376. Epub 2016 May 3. PMID 27140180
- [Background] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Background] Teede H, Deeks A, Moran L. Polycystic ovary syndrome: a complex condition with psychological, reproductive and metabolic manifestations that impacts on health across the lifespan. BMC Med. 2010 Jun 30;8:41. doi: 10.1186/1741-7015-8-41. PMID 20591140